CLINICAL TRIAL: NCT05592496
Title: Bilateral Retromuscular Rectus Sheath Block Catheters Usage for Early Postoperative Analgesia After Laparotomic Gastrectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Riga East Clinical University Hospital (Other Government)
Collaborators: University of Latvia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2022-10-06; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Active Comparator): Patients after laparotomic gastrectomy and musculus rectus sheath block and continuous analgesia with 0,125% bupivacaine solution for 72h
  Interventions: Procedure: Bilateral retromuscular rectus sheath block catheters usage for early postoperative analgesia after laparotomic gastrectomy.; Device: Catheter insertion technique by using special tube t; Procedure: Connection of catheters bilateraly to "easy pump" system,; Diagnostic Test: VAS scale for pain control
- Control group (Placebo Comparator): Patients after laparotomic gastrectomy, musculus rectus sheath block and induction of 0,9% NaCl Solution by using "easy pump" system for 72 h
  Interventions: Procedure: Bilateral retromuscular rectus sheath block catheters usage for early postoperative analgesia after laparotomic gastrectomy.; Device: Catheter insertion technique by using special tube t; Procedure: Connection of catheters bilateraly to "easy pump" system,; Diagnostic Test: VAS scale for pain control

INTERVENTIONS:
Procedure: Bilateral retromuscular rectus sheath block catheters usage for early postoperative analgesia after laparotomic gastrectomy. — After surgery patients in the Block group receives continuous 0.125% (10-12 mg/h) bupivacaine infusion through rectus sheath catheters for 72 h in addition to fentanyl i/v infusion on postoperative day 0, and ketorolac or trimeperidine injection on postoperative day 1-2 if necessery. Patients in the Control group receives NaCl 0,9% infusion and fentanyl i/v infusion on postoperative day 0 and ketorolac or trimeperidine injection on postoperative day 1-2 if necessery Pain intensity is going to be assessed in both groups using 0-100 mm Visual Analog Scale (VAS) at 24, 48 and 72 hour intervals after surgery at rest and during movement (by asking the patient to bend legs). Postoperative complications, hospital stay, comorbidities, the time taken to start walking after the surgery, bowel movements (time until first stool) were all examined.
  Other Names: Catheter insertion technique by using special tube to positionate it in retromuscular space
Device: Catheter insertion technique by using special tube t — By using special tube, it is possible to locate the catheters in retromuscular space, where they are close to cutaneous nervs
Procedure: Connection of catheters bilateraly to "easy pump" system, — Connection of catheters, which are inserted in to retromuscular space, to ensure continuous receiving of Bupivacaine fluid for analgesia. "Easy pump" system provides continous receiving of bupivacaine fluid infusion speed - 5ml per hour
Diagnostic Test: VAS scale for pain control — By using Visual Analog scale of pains, the pain score is fixed

SUMMARY:
In early postoperative period, the occurrence of severe pain after open major upper GI surgery is a significant issue. The study is aimed to access the efficiency of rectus sheet block with continuous bupivacaine infusion catheters into retromuscular space in providing an effective pain relief, decreasing opioid consumption and enhancing postoperative recovery.

DETAILED DESCRIPTION:
This prospective randomised case-control experimental study is being conducted in Riga East University Hospital (Latvia). Patients with total or subtotal open gastrectomy were divided into two groups - half patients in the Block group and half patients in the Control group. In the Block group and control group, retromuscular catheters in the m. rectus abdominis sheath is going to be placed before fascia closure. Catheters will be placed under the direct supervision of a surgeon throughout the operation wound on both sides of the incision.

After surgery patients in the Block group will receive continuous 0.125% (10-12 mg/h) bupivacaine infusion through rectus sheath catheters for 72 h. Additionaly ketorolac or trimeperidine infusion will be performed if VAS of pains more than 30mm. If pains continue, additional opioids will be performed.

Patients in the Control group received 0,9% NaCl solution 72 hours by using the same "easy pump" system, and ketorolac or trimeperidine injection if necessery Pain intensity will be assessed in both groups using 0-100 mm Visual Analog Scale (VAS) at 24, 48 and 72 hour intervals after surgery at rest and during movement (by asking the patient to bend legs). Postoperative complications, hospital stay, comorbidities, the time taken to start walking after the surgery, bowel movements (time until first stool) were all examined.

ELIGIBILITY:
Inclusion Criteria:

* Open Laparotomy and gastrectomy

Exclusion Criteria:

* acute surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 3 days
  Patients will be asked to score their pain in recovery and on days 0,1,2,3 post surgery
Opioid usage after surgery | 3 days
  If the VAS of pains is more than 30mm, after receiving NSAIDs, opioid solution will be performed

SECONDARY OUTCOMES:
Peri-operative analgesic use | 4 days
  Analgesic use intra-operatively and post-operatively for 3 days. This will include strong opioids, paracetamol, NSAIDs, codeine, ketamine, IV lignocaine, tramadol, clonidine and PCA usage post-operatively.
TIme to diet and mobilisation | likely 5 days
  Time to first defecation
Time to discharge | approximately 7 days
  how many days after Surgery
Postoperative complications | approximately 14 days
  all postoperative complications (Clavien Dindo classification)

CONTACTS AND LOCATIONS:
Locations (2):
- Latvia (2):
  - Igors Ivanovs, Riga
  - Riga East Clinical University hospital, Riga

IPD SHARING:
Plan to Share IPD: Undecided